CLINICAL TRIAL: NCT05497206
Title: A Post-Market, Multi-Center, Single Arm Trial on Robotic Instrumentation (ROSA® Hip System) in Patients Undergoing Direct Anterior Total Hip Arthroplasty With Fluoroscopic Guidance
Brief Title: ROSA® Hip System THA PMCF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The data needed for regulatory submissions based on the current pace of the study, will not be available in the foreseeable future.
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMU2021-26TDS
Record Dates: First submitted 2022-02-23; First posted 2022-08-11 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: Osteoarthritis, Hip; Avascular Necrosis of Hip
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Robotic-Assisted THA (Experimental): Consecutive participants will receive THA via the ROSA Hip System.
  Interventions: Device: One of the following hip implants may be used within this arm of the study: G7 Acetabular System, Taperloc Complete System, Avenir and Avenir Complete Systems, and Echo Bi-Metric System

INTERVENTIONS:
Device: One of the following hip implants may be used within this arm of the study: G7 Acetabular System, Taperloc Complete System, Avenir and Avenir Complete Systems, and Echo Bi-Metric System — Total Hip Arthroplasty

SUMMARY:
This study is a Prospective, Multicenter, Single-Arm, Cohort post-market study to evaluate the accuracy of acetabular implant position using the robotic-arm surgical assistant (ROSA® Hip System).

DETAILED DESCRIPTION:
Consecutive patients who meet all of the inclusion criteria and none of the exclusion criteria will be eligible for participation in the study, and will be pre-screened for participation in the informed consent process.

The primary objective of this study is to assess the accuracy of acetabular implant position by evaluating the percentage of participants who are within the range of the Callanan safe zones for Acetabular Inclination (30 - 45 degrees). A patient is considered a success if their intra-operative and/or post-operative full pelvis fluoroscopic or radiographic images show the postoperative acetabular inclination to be within this safe zone range.

Secondary Objectives include the evaluation of safety and efficacy of this system and will include the assessment of common adverse events, physical exam findings, radiologic results, and patient reported outcome measures.

Data collection will occur at the following intervals: Pre-operative, Operative, 3-months, 1-year, and 2-years. Enrollment for the study is anticipated to last approximately 18 months. Allowing for 24 months of follow-up, the total estimated study time to final-patient final-visit will be approximately 42 months.

ELIGIBILITY:
Inclusion:

1. Age 18 - 80 years
2. Body mass index ≤40 (BMI = kg/m2)
3. Patient is willing and able to provide informed consent
4. Patient qualifies for primary THA, via an anterior approach, due to osteoarthritis or avascular necrosis of the hip based on Investigator's clinical judgment
5. Independent of study participation, patient is a candidate and meets the indications and none of the contraindications for use with the ROSA Hip System

Exclusion:

1. Has undergone an orthopaedic procedure of the spine or lower extremity, or is currently participating in a pain management clinical study of any joint, within the last 6 months or planned within the next 6 months
2. Patients receiving simultaneous bilateral hip arthroplasties are excluded from participation in this study; as well as any participants with staged bilateral arthroplasties within 6 months of each other
3. Active infection, sepsis, osteomyelitis
4. Patient is at a high risk for dislocation including those with long-segment spinal fusions (>3 levels) and neuromuscular disorders
5. Inflammatory (rheumatoid or psoriatic arthritis) or post-traumatic arthropathy, or any other degenerative joint disease not consistent with osteoarthritis
6. Would, in the Investigator's opinion, be unwilling or unable to comply with the postoperative follow-up schedule
7. Patient is considered a member of a vulnerable population (pregnant, prisoner, mentally incompetent, etc.)
8. Previous hardware in the proximal femur or acetabulum from a prior orthopaedic procedure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2024-06-05 (Actual); Primary Completion 2024-12-12 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Accuracy of implant position | 90 days
  To evaluate the accuracy of acetabular implant position using the robotic-arm surgical assistant (ROSA® Hip System) (rTHA). Accuracy of acetabular implant position will be assessed by evaluating the percentage of participants who are within the range of the Callanan safe zones for Acetabular Inclination (30 - 45 degrees). A patient is considered a success if their intra-operative and/or post-operative full pelvis fluoroscopic or radiographic images show the postoperative acetabular inclination to be within this safe zone range.

SECONDARY OUTCOMES:
Evaluation of Patient safety | 24 months
  Frequency and incidence of adverse events, serious adverse events, adverse device effects, serious adverse device effects, and unanticipated serious adverse device effects as well as device deficiencies.
Patient Reported Outcome Measure (Oxford Hip Score) | 24 months
  A questionnaire completed by the patient consisting of twelve questions that utilize a 5-point Likert scoring system (0 - 4) resulting in a score ranging from 0 (worst) to 48 (best).
Numeric Pain Rating Scale (NPRS) | 24 months
  An 11-point NPRS is a patient self-completed reported outcome and will be used to assess the current level of pain for the affected hip. On this scale, 0 will indicate no pain and 10 will indicate the worst pain imaginable
Subject Satisfaction | 24 months
  A questionnaire consisting of a single satisfaction question in regard to the subjects hip replacement. Answers will include the following: Very Dissatisfied, Dissatisfied, Neutral, Satisfied, Very Satisfied.
Clinical performance will be assessed with evaluation of range of motion. | 24 months
  Range of motion will be evaluated in a supine position and assess flexion, abduction (in flexion), adduction (in flexion), external rotation (in extension), and internal rotation (in extension). Range of motion will be measured in degrees.
Clinical performance will be assessed with evaluation of stability using the Trendelenburg test. | 24 months
  The test is negative when the hip of the leg that is lifted, will also go up i.e., hiking of hip or the pelvis tilts upwards. The test is positive, when there is a drop of the hip or a downwards tilt of the pelvis. The test is level when the subject presents normal gait and adequate pelvic stability. If the subject is unable to perform the test, this will be noted "unable to perform test".
Clinical performance will be assessed by testing leg length discrepancy. | 24 months
  This will be assessed by (3) categories (legs equal, right short, left short) and discrepancies will be measured in mm or cm.
Physician Radiographic Assessment of Acetabular Cup | 2 Years
  Records acetabular cup inclination (degrees), acetabular cup anteversion (degrees)
Physician Radiographic Assessment of Femoral and Global Offset and Leg Length Discrepancy | 2 Years
  Records femoral offset (mm), global offset (mm), leg length (mm)
Physician Radiographic Assessment of Significant Radiographic Findings | 2 Years
  Records evidence of fracture (y/n), evidence of acetabular migration (y/n), evidence of heterotopic ossification (y/n), or other significant radiographic findings (including the zone it occurs in)

CONTACTS AND LOCATIONS:
Overall Officials: Hillary Overholser, Study Director — Zimmer Biomet
Locations (2):
- United States (2):
  - The Mayo Clinic Jacksonville, Jacksonville, Florida
  - Mosaic Life Care, Saint Joseph, Missouri

IPD SHARING:
Plan to Share IPD: No